CLINICAL TRIAL: NCT05297422
Title: Administration of Ketamine to Branchial Plexus Block Using Axillary Approach : Comparative Study
Brief Title: Axillary Approach to Brachial Plexus Blockade Using Ketamine, Regional Versus Intravenous Administration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Demetra Solomou, Anaesthesiology Resident at KAT and Masters Student at National and Kapodistrian University of Athens, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 877/14-01-2022
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Branchial Plexus Blockade; Anesthesia
Keywords: Axillary Approach; Ketamine; Adjuvant
MeSH Terms: interventions — Ropivacaine; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Active Comparator): Axillary Approach to Brachial Plexus Blockade will be performed using 30ml Ropivacaine 0.5% ,without Ketamine as an adjuvant.
  Interventions: Procedure: Forearm surgey; Drug: Ropivacaine
- Ketamine IV (Active Comparator): Axillary Approach to Brachial Plexus Blockade will be performed using 30ml Ropivacaine 0.5% ,with Ketamine as an adjuvant 30mg intravenously.
  Interventions: Procedure: Forearm surgey; Drug: Ropivacaine; Drug: Ketamine
- Ketamine Regional (Active Comparator): Axillary Approach to Brachial Plexus Blockade will be performed using 30ml Ropivacaine 0.5% ,with Ketamine as an adjuvant 30mg regionally.
  Interventions: Procedure: Forearm surgey; Drug: Ropivacaine; Drug: Ketamine

INTERVENTIONS:
Procedure: Forearm surgey — Microsurgery Clinic , KAT Hospital Athens
Drug: Ropivacaine — Ropivacaine
Drug: Ketamine — Ketamine
  Arms: Ketamine IV; Ketamine Regional

SUMMARY:
The purpose of this study is to assess Ketamine as an adjuvant to Branchial Plexus Blockade.

DETAILED DESCRIPTION:
After being informed about the study, patients giving written informed consent will undergo anaesthesia using the Ultrasound Guided Axillary Approach to Brachial Plexus Blockade, in order to undergo forearm surgery. The purpose of this study is to assess whether Ketamine as an adjuvant lengthens sensory and motor blockade and whether it has an effect on "rebound pain" when the anaesthetic effect fades. Therefore the study will compare intravenous, regional and no administration of Ketamine as an adjuvant to Branchial Plexus Blockade. Patients will be asked to fill in a Pain VAS (Visual Analog Scale) for 24 hours following the intervention, in order to assess effectiveness of each anaesthetic method. Side effects, onset time, motor blockade score and rescue dose are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-35
* ASA score I, II, III

Exclusion Criteria:

* Mental disorder
* Peripheral neuropathy
* Severe hepatic or renal disease
* Gastrointestinal bleeding history

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
VAS (Visual Analog Scale) over 24 hours following intervention | 24 hours
  VAS scale is expressed in integer numbers ranging from 0-10, where 0=no pain, 10= excruciating pain.

SECONDARY OUTCOMES:
Side Effects | 24 hours
  Dizziness, nausea, vomiting, paraesthesia
Motor Blockade Score | 24 hours
  0=complete paralysis, 1=partial paralysis, 2=no paralysis
Anesthesia Onset time | 24 hours
  Time from removal of needle to final motor and sensory blockade result
Rescue Dose | 24 hours
  Tramadol 100mg intravenously administered only to patients who claim to be in strong pain within the 24 hours after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Xanthos, Professor, Study Director — National Kapodistrian University of Athens
Locations (1):
- National and Kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Plan under study
Supporting Information: Study Protocol
Time Frame: June 2023

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/10781465/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4260270/